CLINICAL TRIAL: NCT05357924
Title: Evaluating Ovarian Reserve After Conventional Laparoscopy Versus Robotic Surgery for Bilateral Endometrioma: a Randomized Controlled Trial.
Brief Title: Evaluating Ovarian Reserve After Conventional Laparoscopy Versus Robotic Surgery for Bilateral Endometrioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christine Bekos, Principan Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMH robotic LSK
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Ovarian Endometrioma; Ovarian Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- robotic-assisted laparoscopy (Active Comparator): The robotic-assisted resection of endometriosis will be performed using the da Vinci Surgical System Si (Intuitive Surgical) using up to five ports as needed. An umbilical port was placed for the laparoscope (10/12 mm), a 5-mm port for the assistant, and two to three ports (5/8 mm) for the robotic arms.
  Interventions: Procedure: robotic-assisted laparoscopy
- conventional laparoscopy (Active Comparator): Laparoscopic-assisted cystectomy of endometrioma will be performed using up to four 5-mm ports, including an umbilical port and additional ports as dictated by each individual surgery.
  Interventions: Procedure: Conventional laparoscopy

INTERVENTIONS:
Procedure: robotic-assisted laparoscopy — Superficial and deep endometriosis resection will be performed in the usual standard fashion. All superficial lesions suspicious for endometriosis (pigmented and nonpigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy will be performed for endometriomas. Additional procedures are performed as needed to completely resect all endometriosis lesions. The fascia of any port ≥10 mm will be reapproximated. Cystoscopy will be performed when deemed appropriate by the surgeon. If bowel resection and re-anastomosis is necessary this will be performed together with a General Surgeon.
  Other Names: DaVinci laparoscopy
  Arms: robotic-assisted laparoscopy
Procedure: Conventional laparoscopy — Superficial and deep endometriosis resection will be performed in the usual standard fashion. All superficial lesions suspicious for endometriosis (pigmented and nonpigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy will be performed for endometriomas. Additional procedures are performed as needed to completely resect all endometriosis lesions. The fascia of any port ≥10 mm will be reapproximated. Cystoscopy will be performed when deemed appropriate by the surgeon. If bowel resection and re-anastomosis is necessary this will be performed together with a General Surgeon.
  Arms: conventional laparoscopy

SUMMARY:
The aim of this study is to perform a randomized study investigating AMH recovery comparing robot-assisted laparoscopy and conventional laparoscopy in patients with bilateral ovarian endometrioma. It is hypothesized that in patients with endometriomas, a robot-assisted approach may provide improved instrument navigation resulting in more precise dissection and therefore removal of less healthy ovarian tissue compared to conventional laparoscopy. AMH is the most widely used parameter for predicting functional ovarian reserve. Postoperative AMH levels were associated with the number of follicles in specimens due to the removal of ovarian cortex during surgery . Furthermore, the reduction in AMH level after surgery is higher in bilateral endometrioma.

The investigators hypothesize, on the basis of Lee at al., 2020, that patients with bilateral endometrioma will have significantly higher AMH levels 6 months after robot-assisted laparoscopy than patients who were treated with conventional laparoscopy.

Therefore, the primary outcome is postoperative serum AMH level recovery in patients undergoing conventional laparoscopy versus robot-assisted laparoscopy.

Aims: The aim of this study is to investigate postoperative differences in ovarian reserve differing between robot-assisted laparoscopy compared to conventional laparoscopy in patients with bilaterial ovarian endometrioma by comparing serum AMH (sAMH) level recovery.

Study population: The study population will consist of women aged between 18 and 45 years who are referred to our gynecologic outpatient clinic due to bilateral endometrioma. Women with an indication for surgery can be included in this trial.

Methods: Laparoscopic-assisted resection of endometriosis will be performed using up to four 5-mm ports, including an umbilical port and additional ports as dictated by each individual surgery. The robotic-assisted resection of endometriosis will be performed using the da Vinci Surgical System Si (Intuitive Surgical) using up to five ports as needed. Superficial and deep endometriosis resection will be performed in the usual standard fashion. Histological confirmation of endometriosis will be performed. The primary outcome is postoperative serum AMH (sAMH) level recovery. This will be evaluated 6 months after surgery.

DETAILED DESCRIPTION:
Experimental Plan

Study design This trial is a prospective, randomized-controlled study investigating postoperative differences in ovarian reserve differing between robot-assisted laparoscopy compared to conventional laparoscopy in patients with bilaterial ovarian endometrioma by comparing serum AMH (sAMH) level recovery. Postoperative follow-up will take place after 6 months. All women referred to our department for endometrioma will undergo clinical examination by a senior surgeon experienced in endometriosis as well as ultrasound. All patients with bilateral endometrioma will be included. Complementary examinations, such as cystoscopy or renal sonography will be performed in women with suspected involvement of urinary tract.

In women with pregnancy intention and endometrioma, an exhaustive assessment of the disease will systematically be performed before deciding between primary surgery and primary assisted reproductive techniques.

Gynecological examination will be performed at each visit. Ovarian reserve will be evaluated using antral follicle count (AFC) via transvaginal sonography, anti-Mullerian hormone (AMH), follicle-stimulating hormone (FSH) and luteinizing hormone (LH) levels and ovarian volume.

Follicle number will be evaluated by pathologists in the histologic tissue sections.

Furthermore, subjective outcome will be assessed with standardized questionnaires.

Study setting This study will be conducted at the gynecologic outpatient clinic (Division of General Gynecology and Gynecologic Oncology, Department of Obstetrics and Gynecology, Medical University of Vienna). Enrollment, treatment and data collection will be standardized by all sites according to the approved study protocol.

Participants and recruitment The study population will consist of women aged between 18 and 45 years who are referred to our gynecologic outpatient clinic due to endometrioma. Women with bilateral endometrioma and an indication for surgery can be included in this trial.

Intervention Laparoscopic-assisted cystectomy of endometrioma will be performed using up to four 5-mm ports, including an umbilical port and additional ports as dictated by each individual surgery. The robotic-assisted resection of endometriosis will be performed using the da Vinci Surgical System Si (Intuitive Surgical) using up to five ports as needed. An umbilical port was placed for the laparoscope (10/12 mm), a 5-mm port for the assistant, and two or three ports (5/8 mm) for the robotic arms. Superficial and deep endometriosis resection will be performed in the usual standard fashion. All superficial lesions suspicious for endometriosis (pigmented and nonpigmented) will be completely resected until non-diseased peritoneal margins are visualized around the defect; all deep lesions suspicious for endometriosis will be completely resected until non-diseased margins are visualized in the tissue surrounding the defect. Cystectomy will be performed for endometriomas. Additional procedures are performed as needed to completely resect all endometriosis lesions. The fascia of any port ≥10 mm will be reapproximated. A cystoscopy will be performed when deemed appropriate by the surgeon. If bowel resection and re-anastomosis are necessary this will be performed together with a General Surgeon.

Participating surgeons will be defined as high-volume surgeons in endometriosis surgery and will also be part of the endometriosis core team.

Histological confirmation of endometriosis will be performed.

Postoperative Management: The patients are instructed to rest for 2 weeks after the operation (not to work, do sport, do the cleaning, and carry more than five kilos). They are allowed to return to work after 2 weeks and to take part in sports or have intercourse after 6 weeks. Follow-up visits are scheduled after 6 months in our outpatient clinic due to our study protocol.

For the postoperative medical treatment of endometriosis, combined oral contraceptive, a GnRH agonist or Dienogest will be administered to all patients who do not desire pregnancy. Patients desiring pregnancy will either be advised to attempt spontaneous conception or will be sent to our in-house ART department depending on their age, disease extent, preoperative AMH levels and male factors.

Data collection At baseline, the following data will be collected: demographics and medical history data (age, body mass index, parity, menopausal and hormone therapy status, current smoking, previous adnexal surgery, and medical comorbidities (diabetes mellitus, connective tissue disorders)). Previous endometriosis-specific treatments and responses will be assessed. Patients will be asked to complete the Endometriosis Health Profile (EHP) EHP-30 25. A gynecological examination will be performed at each visit. Ovarian reserve will be evaluated using antral follicle count (AFC), anti-Mullerian hormone (AMH), follicle-stimulating hormone (FSH), and luteinizing hormone (LH) levels, and ovarian volume.

Preferentially, LH and FSH will be evaluated in the first 2 to 5 days of the menstrual cycle.

The patients will be asked to rate their satisfaction with the appearance of their scars on a 10-point Likert scale (with 1 being very unsatisfied and 10 being very satisfied).

ELIGIBILITY:
Inclusion Criteria:

* Bilateral endometrioma
* Surgical endometriosis resection is planned
* sAMH > 1.0 ng/ml

Exclusion Criteria:

* History of malignant diseases
* History of adnexal surgery
* Subject is unable or unwilling to participate
* Postmenopausal women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum AMH (sAMH) from baseline to 6 months after the operation | 6 months after the operation
  postoperative sAMH (6 months after the operation) compared to preoperative sAMH

SECONDARY OUTCOMES:
Change in antral follicle count (AFC) from baseline to 6 months after the operation | 6 months after the operation
  antral follicle count (AFC) measured via transvaginal sonography
change in ovarian volume from baseline to 6 months after the operation | 6 months after the operation
  ovarian volume measured via transvaginal sonography (preoperative ovarian volume - endometrioma volume versus postoperative ovarian volume)
change in follicle-stimulating hormone (FSH) and luteinizing hormone (LH) from baseline to 6 months after the operation | 6 months after the operation
  postoperative FSH and LH(6 months after the operation) compared to preoperative FSH and LH (both times measured within the first 2-5 days of menstrual cycle)
rate of intraoperative adverse events | 1 day
  rate of intraoperative adverse events (bladder injury, bowel injury, ureteral obstruction, massive bleeding)
rate of postoperative adverse events | 4 weeks
  rate of postoperative adverse events related to surgery (classified using Clavien Dindo classification)
operation time | 1 day
  operation time in minutes
length of hospitalization (following the operation) | 2 weeks
  length of hospitalization in days
blood loss | 1 day
  change of hemoglobin levels 24 hours after surgery
laparotomic conversion rate | 1 day
  laparotomic conversion rate
follicle number in the histologic tissue sections | 1 day
  follicle number in the histologic tissue sections
change of the Endometriosis Health Profile (EHP) EHP-30 from baseline to 6 months after the operation | 6 months after the operation
  questionnaires: the Endometriosis Health Profile (EHP) EHP-30 (preoperative versus 6 months after the operation
10-point Likert scale for cosmetic satisfaction | 6 months after the operation
  questionnaires: 10-point Likert scale for cosmetic satisfaction
Disease recurrence rate up to 12 months after surgery | 12 months after the operation
  Endometriosis recurrence can have different levels: symptoms recurrence based on patient history (VAS pain score ≥ 5), but no proof of recurrence by imaging and/or surgery; endometriosis recurrence based on non-invasive imaging in patients with or without symptoms; recurrence of histologically proven endometriosis: when the patient is re-operated, endometriosis is visually observed and confirmed histologically.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Wenzl, Study Director — Medical University of Vienna, Department of Obstetrics and Gynecology
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No